CLINICAL TRIAL: NCT05710744
Title: Mitigating Racial Disparities in Shared Decision Making in the Intensive Care Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00111530; 1K23HL164968-01 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Health Care Disparities
Keywords: Intensive Care Unit; Racial Disparities in Healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Members of patients in the ICU (No Intervention): Family members will join routine meetings with the physicians treating with their critically ill loved ones.
- ICU Physicians (Other): Physicians will view a tip sheet containing information about best practices of shared decision making with diverse individuals. Physicians will then conduct routine meetings with families of patients with acute respiratory failure.
  Interventions: Behavioral: Shared decision making tip sheet

INTERVENTIONS:
Behavioral: Shared decision making tip sheet — Physicians will view tip sheets containing best practices for shared decision making with diverse families.
  Arms: ICU Physicians

SUMMARY:
This is a non randomized pilot trial aimed to:

Test the feasibility of an intervention to support intensive care unit clinicians in conducting shared decision making conversations with families of patients with acute respiratory failure. The goal of this intervention is to mitigate racial disparities in shared decision making.

DETAILED DESCRIPTION:
The care of critically ill patients with acute respiratory failure involves life-or-death decisions. Ideally, intensive care unit (ICU) clinicians should include patients or their families in shared decision making, which promotes goal-concordant care (i.e., care aligned with patients' preferences), reduces psychological distress for both families and clinicians, and shortens ICU length of stay. However, racial disparities have been documented in shared decision making and associated outcomes. In outpatient settings, clinicians treat Black patients differently from White patients, providing fewer treatment options, less prognostic information, and less emotional support, and making assumptions about rather than eliciting patient preferences. Disparities in shared decision making are likely to be amplified in the ICU because clinicians often do not have long-standing relationships with patients or families, and decisions are complex, emotional, and time-pressured. Yet, no interventions currently exist to address racial disparities in shared decision making about acute respiratory failure. This research will directly fill this gap.

ELIGIBILITY:
Physician inclusion criterion:

- ICU attending physician with at least 6 weeks of clinical service time in the 12 months preceding and following enrollment

Physician exclusion criterion:

- Board certified in palliative care medicine

Patient inclusion criteria:

* Admitted to the ICU
* Being treated by a study physician currently and at least for the next 48 hours
* ≥ 18 years of age upon admission to hospital
* Mechanically ventilated ≥ 4 days

Patient exclusion criterion:

* Tracheostomy tube present or decision to pursue tracheostomy within next 7 days
* Has decision making capacity as assessed by medical team
* Extubation planned or death anticipated in next 24 hours
* Patients who are prisoners or are pregnant
* Awaiting organ transplantation during this hospitalization
* Acute respiratory failure due to progression of chronic neuromuscular disease
* No family decision maker available

Family member inclusion criteria:

* Identified by medical team as person most involved in medical decision making for the patient
* Confirmed to be patient's legally authorized representative
* Self-identifies as non-Hispanic, Black or White
* ≥ 18 years of age at time of consent
* Confirms conversational fluency in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability as measured by single Likert-scaled item completed by physicians | within 96 hours of signing study consent
  Likert-scaled single item, ranging from 1 (not acceptable) to 5 (completely acceptable)
Demand for the intervention measured by the proportion of physicians who viewed the intervention | within 96 hours of signing study consent
  Percentage of physicians who viewed intervention by email "read" receipts, range 0 to 100%
Fidelity to intervention measured by proportion of tip sheet phrases used by physicians | within 96 hours of signing study consent
  Proportion of tip sheet phrases used in family meeting as determined by review of audio-recorded family meeting, range 0 to 100%
Practicality as measured by proportion of screen eligible participants enrolled per month | through study completion, up to 1 year
  Proportion screen eligible enrolled/month based on review of study logs, range 0 to 100%
Practicality as measured by time to complete physician or family surveys | within 96 hours of signing study consent
  Time to complete physician or family surveys as measured by review of study logs, range 0 to 60 minutes
Practicality as measured by dropout rate from study | through study completion, up to 1 year
  Dropout rate as ascertained by review of study logs, range 0 to 100%

SECONDARY OUTCOMES:
Decisional regret among families, measured by Decision Regret Scale | within 96 hours of signing study consent
  Decision Regret Scale, range 5 (low regret) to 25 (high regret)
Psychological distress among families, measured by Impact of Events Revised scale | within 96 hours of signing study consent
  Impact of Events revised scale, range 0 (low stress) to 88 (extreme stress)
Psychological distress among physicians, measured by moral distress scale | within 96 hours of signing study consent
  Moral distress scale, range 0 (low distress) to 84 (extreme distress)
Components of shared decision making, as measured by content analysis of family meeting recordings | through study completion, up to 1 year
  A qualitative data analysis of transcripts from family-physician meetings using 14-item shared decision making framework from PMID 20642362, range 0 (poor shared decision making) to 14 (ideal shared decision making)
Decisional conflict among families, measured by Decisional Conflict Scale | within 96 hours of signing study consent
  Decisional Conflict Scale, range 0 (low conflict) to 64 (high conflict)
ICU utilization among patients, as measured by length of stay | through study completion, up to 1 year
  ICU length of stay ascertained from electronic medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Deepshikha Ashana, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No